CLINICAL TRIAL: NCT00217113
Title: An Intervention to Preserve Functional Status and Independence Among Community Dwelling Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Minnesota Department of Human Services (Other Government); Elder Network (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1752-05
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Elderly

INTERVENTIONS:
Behavioral: Geriatric home visit and Action Plan

SUMMARY:
This is a study aimed at identifying Olmsted County senior citizens who are at risk for vulnerability. Those elders who screen "affirmatively" for vulnerability will be offered participation in a pilot intervention aimed at keeping seniors independent in the community. This intervention consists of a comprehensive geriatric home visit and the development of an individualized action plan aimed at preservation of function and independence. Participants will be followed for several months after their baseline assessment to evaluate implementation of recommendations.

ELIGIBILITY:
Age 65 or older Olmsted County Resident Able to provide own consent English speaking or with available translator

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Change in VES-13 score (Pre/Post)
Implementation of "Action Plan" Recommendations
Frailty Domain Scores

SECONDARY OUTCOMES:
Hospitalization and Nursing home admissions

CONTACTS AND LOCATIONS:
Overall Officials: Ericka E. Tung, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States